CLINICAL TRIAL: NCT03094650
Title: The Use of Immersive Virtual Reality for Upper Limb Neurorehabilitation in Stroke Survivors
Brief Title: Immersive Virtual Reality for Stroke Motor Rehabilitation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mindmaze SA (Industry)
Collaborators: Ecole Polytechnique Fédérale de Lausanne (Other); Clinique Romande de Readaptation (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Purpose: Treatment
Other Study IDs: MindMaze-2015-CT01
Record Dates: First submitted 2017-03-14; First posted 2017-03-29 (Actual); Last update posted 2017-03-29 (Actual); Status verified 2017-03

CONDITIONS: Chronic Stroke; Motor Disorders
Keywords: stroke; neurorehabilitation; virtual reality; rehabilitation dose; motor rehabilitation
MeSH Terms: conditions — Motor Disorders; Stroke

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MindMotion PRO (Experimental): The training sessions consist of virtual reality based rehabilitation exercises using the MindMotion PRO device.
  Interventions: Device: MindMotion PRO

INTERVENTIONS:
Device: MindMotion PRO — Patients will receive five weeks of therapy with 2 sessions (minimum) per week lasting for 45-60 minutes each minimum. The training sessions are based on the MindMotion PRO's virtual reality exercises.

SUMMARY:
The present study aims at investigating (i) the feasibility in chronic stroke of using a dedicated virtual reality (VR) based system that embeds real-time 3D motion capture and embodied visual feedback to deliver functional exercises designed for training of impaired upper limb motor skills, (ii) whether chronic stroke survivors improve in functional outcomes in the upper limb when exposed to intensive VR-based therapy, and (iii) safety and tolerance to such a technology. The investigators hypothesize that intensive VR-based rehabilitation may lead to high rehabilitation doses and functional improvement in chronic stroke.

ELIGIBILITY:
Inclusion Criteria:

* Ischemic or hemorrhagic minor-to-moderate (0<NIHSS<16) stroke with hemiparesis and experiencing arm motor difficulties
* At least 6 months after stroke incident
* Maximum 4 on the Medical Research Council Scale (MRCS) for shoulder elevation and elbow flexion/extension
* 18 years and older
* First ever stroke

Exclusion Criteria:

* Participating in another movement treatment study at the time of the present study
* Severe cognitive impairment (Mini Mental Status Examination score < 18 points)
* Orthopedic impairment or visual disorders limiting the treatment
* Unable to give informed consent form
* Risk of epileptic seizures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2015-02 (Actual); Primary Completion 2015-10 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Rehabilitation dose: goal-directed movements (i.e. number of intended movements to achieve a task) | 5 weeks
  Rehabilitation dose: goal-directed movements (i.e. number of intended movements to achieve a task)
Training intensity: number of goal-directed movements per minute of effective training time. | 5 weeks
  Training intensity: number of goal-directed movements per minute of effective training time.
Change in Upper limb function assessed with Fugl-Meyer Assessment for Upper Extremity (FMA-UE) | At baseline, 5 weeks (post intervention) and 9 weeks (follow-up)
  Fugl-Meyer Assessment for Upper Extremity (FMA-UE)

SECONDARY OUTCOMES:
Change in Functional Independence Measure (FIM) | At baseline, 5 weeks (post intervention) and 9 weeks (follow-up)
Change in kinematic metrics/goniometry (active range of motion). | At baseline, 5 weeks (post intervention) and 9 weeks (follow-up)
Change in Modified Medical Research Council Scale (mMRCS) | At baseline, 5 weeks (post intervention) and 9 weeks (follow-up)
Change in Visual Analog Scale (VAS) for Pain | At baseline, 5 weeks (post intervention) and 9 weeks (follow-up)
Safety and Acceptance of Technology assessed with a questionnaire | 5 weeks
  Participants will answer a questionnaire to evaluate following aspects:
  * Tolerance to VR intervention
  * Adverse event monitoring
  * Self-evaluation
  * Acceptance of technology
  * Motivation

CONTACTS AND LOCATIONS:
Locations (1):
- Center for Neuroprosthetics-Valais (EPFL) at Clinique Romande de Réadaptation, Sion, Valais, Switzerland

REFERENCES:
- [Derived] Perez-Marcos D, Chevalley O, Schmidlin T, Garipelli G, Serino A, Vuadens P, Tadi T, Blanke O, Millan JDR. Increasing upper limb training intensity in chronic stroke using embodied virtual reality: a pilot study. J Neuroeng Rehabil. 2017 Nov 17;14(1):119. doi: 10.1186/s12984-017-0328-9. PMID 29149855